CLINICAL TRIAL: NCT04541121
Title: Effects of 3D Ultrasonography and 3D Printed Images on Maternal-fetal Attachment and Its Correlation With Overall Smoking Within Pregnancy and Smoking Cessation
Brief Title: 3D Maternal Fetal Attachment and Smoking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2001287
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Maternal-Fetal Relations; Maternal Behavior

STUDY DESIGN:
Intervention Model Description: 3D ultrasound and picture of ultrasound or 3D ultrasound and printed model of fetal face
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed model (Experimental): Mother is given 3D printed model of fetus' face
  Interventions: Behavioral: 3D printed model
- Placebo (Placebo Comparator): Mother is given printed picture of 3D ultrasound of fetus
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: 3D printed model — Mother is given 3D printed model of fetus' face
  Other Names: Mother is given 3D printed model of fetus' face
  Arms: 3D printed model
Behavioral: Placebo — Mother is given a picture of 3D ultrasound of fetus
  Arms: Placebo

SUMMARY:
To determine whether 3D models of fetus' face created from 3D ultrasound will increase maternal attachment and aid in smoking cessation. Half of participants will receive 3D model and half will receive a picture of 3D ultrasound of their baby

ELIGIBILITY:
Inclusion Criteria:

* Age - Female 19-45 years of age
* Fluent in English
* Currently smoking cigarettes
* Currently pregnant (between 21- and 36-weeks' gestation)
* Have normal 20-week ultrasound

Exclusion Criteria:

* Having received more than 3 ultrasounds prior to study
* Medical need for additional ultrasounds
* Multiple fetuses
* > 31 weeks gestation
* Does not smoke cigarettes
* Is not fluent in English

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women currently pregnant (between 21- and 36-weeks' gestation)
Enrollment: 96 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal Antenatal Attachment Scale (MAAS) | 5 minutes
  The MAAS is a 19 item questionnaire measuring maternal-fetal attachment. Each item has five answer choices scored from 1 low attachment to 5 high attachment such that the total score ranges from 19 to 95. The measure also includes two subscales: (1) Quality of Attachment has 10 items with a range of 10-50 and measures the quality of the mother's attachment to her fetus. (2) Time measures the time spent in attachment mode (or intensity of preoccupation) and consists of 8 items for a range of 8 to 40. (for clarity one item included in the total score is not included in either subscale.)
The Timeline Follow Back (TLFB): | 10 minutes
  This semi-structured interview utilizes a calendar to aid in participants' recall of smoking throughout pregnancy. The TLFB method is the preferred approach to measure substance use and has shown reliability when used for pregnant women in previous studies
Salivary cotinine | 5 minutes
  Cotinine is a stable nicotine metabolite produced by the liver. This is to test amount mother has smoked.

CONTACTS AND LOCATIONS:
Overall Officials: John Cote, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cote JJ, Cote RD, Dilsaver DB, Massey SH, Doehrman P, Cote BP, Kilzer R, Badura-Brack AS. Effects of 3D ultrasonography and 3D printed images on maternal-fetal attachment and its correlation with overall smoking within pregnancy: a pilot study. 3D Print Med. 2024 Oct 30;10(1):35. doi: 10.1186/s41205-024-00238-7. PMID 39475978